CLINICAL TRIAL: NCT02794545
Title: Kaohsiung Medical University Chung-Ho Memorial Hospital Tropical Medicine Center
Brief Title: Functional Cure Study of HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KMUHIRB-20140058
Record Dates: First submitted 2016-03-26; First posted 2016-06-09 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2016-09

CONDITIONS: HIV
MeSH Terms: interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recent infection patient (Experimental): The patient who infected with HIV-1 and screened out by P24 ELISA, and they would receives early cART course.
  Interventions: Procedure: cART course

INTERVENTIONS:
Procedure: cART course — The investigators would start regular cART course immediately for early infection patients to achieve functional cure.
  Other Names: HAART

SUMMARY:
Although combination antiretroviral therapy (cART) can significantly reduce morbidity and mortality, it still fails to eradicate HIV. Given the difficulty for eradication of HIV, functional cure is more likely to achieve the goal. In recent breakthrough scientific reports, there already existed several examples of HIV-infected cases achieving the status of functional cure only through early administration of cART in newborns or early infected cases. From Taiwan centers for disease control (CDC) reports and our clinical experiences, more and more young men got HIV infection and the most important finding is the investigators can find some of them are newly infected, let's say, within six months.

DETAILED DESCRIPTION:
This study targets on this newly HIV- infected cohort and urging them to receive cART in order to achieve the possible status of HIV function cure. After 3~5 years period of treatment, cART will be discontinued after laboratory evaluation and functional cure is anticipated. These patients can achieve good life quality. In addition to elimination of the risk for HIV transmission, the cART expense of the government can be reduced on the large scale. The core of this study aims at setting up a precise and standard laboratory methodology for detecting the newly infected cases and predicting the time to stop cART. Once these assay methods are well established, they can be widely applied to assess the previous cases with long term cART for the prediction of the appropriate time to stop cART.

Thru the conventional HIV tests (within the sero-conversion stage), the detection rate of early infection is only 5-10 %. Therefore it is very desperately important to develop more tools for the diagnosis of early infection.

In addition to the standard method for detecting HIV infection, the investigators will use the HIV p24 Ag test and detuned Enzyme-linked Immunoblotting assay (EIA) assay for detecting early infection. For naïve patients, the investigators will also check the resistance testing for antiretroviral drugs in order to adjust and choose the susceptible cART for the patients. During the cART period, the investigators will follow up these patients for checking quantity of HIV RNA and proviral DNA (HIV DNA) from Peripheral blood mononuclear cell (PBMCs) in their blood. After three to five years of cART, if their HIV RNA is not detected and HIV DNA is very low, the investigators will draw the blood from the patients to isolate the Cluster of Differentiation 4 (CD4) receptors + T cells and co-cultivated with PBMCs from the healthy cohorts to evaluate the existence of HIV infectivity or not in the cART treated cases. If there is no infectivity, the investigators will stop cART. After stopping cART, the investigators will follow up these cases every six months till at least two years to check their HIV antibody, HIV RNA and HIV DNA from PBMCs to observe whether HIV recurrence occurs to them.

ELIGIBILITY:
Inclusion Criteria:

1. HIV
2. Age over 20 years old to 35 years old.

Exclusion Criteria:

1. Refuse to accept cases HAART
2. Interruption of HAART cases during treatment.
3. Can not rule taking HAART drugs, leading to treatment failure cases.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
In ELISA format test cases contain the plasma p24 Ag | 3 to 5 years
  Test cases contain the plasma p24 antigen and Detuned assay for early to tell whether a dye.

SECONDARY OUTCOMES:
Monitoring of functional cure | every six months till at least two years
  After three to five years of cART, if the subjects's HIV RNA is not detected and HIV DNA is very low, the investigators would draw the blood from the subjects to isolate the CD4 + T cells and co-cultivated with PBMCs from the healthy cohorts to evaluate the existence of HIV infectivity or not in the subjects. If there is no infectivity, the investigators would stop subjects's cART course.After stopping cART, the investigators would follow up these subjects every six months till at least two years to check their HIV antibody, HIV RNA and HIV DNA from PBMCs to observe whether HIV recurrence occurs to them.

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Jin Tsai, PhD, Principal Investigator — Tropical Medicine Center (TMC), Kaohsiung Medicine University Hospital (KMUH)
Locations (1):
- Kaohsiung medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided